CLINICAL TRIAL: NCT02261545
Title: The Effect of n-3 Fatty Acid Supplementation on the Expression of Sirt-1, Adiponectin Receptor 1 (AdipoR1) & Adiponectin Receptor 2 (AdipoR2) Genes of PBMC and Circulatory Levels of Resistin,Monocyte Chemotactic Protein (MCP-1) and Adiponectin of type2 Diabetes Patient
Brief Title: The Effect of n-3 Fatty Acid Supplementation on Serum Levels, and Gene Expression of type2 Diabetes Patient
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Tehran University of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 25367
Record Dates: First submitted 2014-10-07; First posted 2014-10-10 (Estimated); Last update posted 2015-11-18 (Estimated); Status verified 2015-11

CONDITIONS: Diabetes Mellitus Type II
Keywords: n-3 fatty acid; Sirt-1; AdipoR1; AdipoR2; MCP-1; Adiponectin; Resistin; T2DM
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Fatty Acids, Omega-3; Docosahexaenoic Acids

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- n-3 Fatty Acid Supplemetation (Active Comparator): patients with Type II Diabetes who receive 3 cap omega3, 3 times a day, for 10 weeks.
  Interventions: Dietary Supplement: n-3 Fatty Acid
- Placebo (Placebo Comparator): patients with Type II Diabetes who receive 3 cap of placebo/ for 10 weeks.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: n-3 Fatty Acid — n-3 Fatty Acid supplement, 3 × 1000 mg softgel daily (2700 mg EPA+DHA per day), 3 times a day, for 10 weeks.
  Other Names: omega-3; n-3 PUFA
  Arms: n-3 Fatty Acid Supplemetation
Dietary Supplement: Placebo — 3 cap 1 g Placebo(paraffin) per day for 10 weeks. Control Group: n-3 Fatty Acid placebo softgel (Containing 3 g edible paraffin oil), 3 × 1000 mg softgel daily (3 g per day), 3 times a day, for 10 weeks.
  Arms: Placebo

SUMMARY:
The aim of this study is to determine the effects of supplementation with n-3 fatty acid or placebo for 10 weeks on the expression of Sirt-1, AdipoR1 & AdipoR2 genes in the peripheral blood mononuclear cell (PBMC) and circulatory levels of Resistin, MCP-1 and Adiponectin of type2 diabetes patient

DETAILED DESCRIPTION:
The aim of this study is to determine of the effects of supplementation with n-3 fatty acid or placebo for 10 weeks on the expression of Sirt-1, AdipoR1(adiponectin receptor 1) & AdipoR2 (adiponectin receptor 2) genes in the peripheral blood mononuclear cell (PBMC) and circulatory levels of Resistin, MCP-1 (Monocyte Chemoattractant Protein-1) and Adiponectin of type2 diabetes patient. In this randomized, double-blind clinical trial, placebo-controlled, 88 men and women with type 2 diabetes are enrolled in the study from the Iranian Diabetes Association. After signing informed consent all individuals complete a general information form , 24-hour food recall for 3 days and beck depression questionnaire will be taken from the participants at the beginning and the end of the study. Selected samples are randomly classified into 2 blocks of groups receiving supplement and placebo. The supplement group, will receive mg 1800mg EPA(Eicosapentaenoic acid ) & 900mg DHA( docosahexaenoic acid) (total=2700mg) for 10 weeks and the placebo group will also receive placebo (containing 2700 mg of edible paraffin) (similar in terms of color, shape and size). Patients are recommended to sustain their diets and medication dose (s) during the study and also advised to maintain a constant level of physical activity. Blood samples will be collected after 12 hours fasting and anthropometric variables, biochemical parameters, target gene expression and physical activity before and after the trial will be measured

ELIGIBILITY:
Inclusion Criteria:

* willingness to participation,
* diabetic patients 30- 60 years old,
* body mass index in the range 25-40,
* avoidance of dietary supplements,
* vitamins and herbal products at least 3 months before and throughout the intervention

Exclusion Criteria:

* people who have used n-3 Fatty Acid Supplementation in last 3 months,
* having chronic renal disease ,
* GI disease,
* Hepatobiliary diseases,
* hematological disorders,
* hypo- or hyperthyroidism,
* type 1 diabetes,
* treatment with orlistat or sibutramine for weight loss,
* pregnancy and lactation,
* treatment with insulin or Thiazolidinediones.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2014-09; Primary Completion 2016-01 (Estimated); Study Completion 2016-02 (Estimated)

PRIMARY OUTCOMES:
Serum Fasting Blood Sugar(FBS) | Change from baseline at 10 weeks

SECONDARY OUTCOMES:
Serum Insulin | Change from baseline at 10 weeks
Serum HbA1C | Change from baseline at 10 weeks
Serum Resistin | Change from baseline at 10 weeks
Serum adiponectin | Change from baseline at 10 weeks
Serum mcp-1 | Change from baseline at 10 weeks
Gene Expression of AdipoR1 | Change from baseline at 10 weeks
Gene Expression of AdipoR2 | Change from baseline at 10 weeks
Gene Expression of Sirt-1 | Change from baseline at 10 weeks
Beck depression score | Change from baseline at 10 weeks
Serum cholesterol | Change from baseline at 10 weeks
Serum LDL cholesterol | Change from baseline at 10 weeks
Serum TG | Change from baseline at 10 weeks
Serum HDL cholesterol | Change from baseline at 10 weeks

REFERENCES:
- [Derived] Mazaherioun M, Saedisomeolia A, Javanbakht MH, Koohdani F, Zarei M, Ansari S, Khoshkhoo Bazargani F, Djalali M. Long Chain n-3 Fatty Acids Improve Depression Syndrome in Type 2 Diabetes Mellitus. Iran J Public Health. 2018 Apr;47(4):575-583. PMID 29900143